CLINICAL TRIAL: NCT03307759
Title: Sequencing of Stereotactic Ablative Body Radiotherapy in Combination With PD-1 Blockade Using Pembrolizumab in Metastatic Non-Small Cell Lung Carcinoma
Acronym: SABRseq
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow patient accrual
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SABRseq
Record Dates: First submitted 2017-10-06; First posted 2017-10-12 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Radiotherapy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SABR plus pembrolizumab (Active Comparator): SABR followed by pembrolizumab
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy (SABR)
- Pembrolizumab plus SABR (Active Comparator): Pembrolizumab followed by SABR after cycle 1
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy (SABR)

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab
Radiation: Radiotherapy (SABR) — Radiotherapy

SUMMARY:
This investigator driven Phase Ib study will examine the safety, efficacy and biological effects of two schedules of pembrolizumab, an antibody targeted against anti-programmed cell death 1 (PD-1), which will be given either before or after stereotactic ablative body radiotherapy (SABR) for metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent for the trial.
2. Be ≥ 18 years of age on day of signing informed consent.
3. Have at least one lesion not planned for SABR that is measurable disease based on RECIST 1.1.
4. Patients must have a histologically or cytologically confirmed metastatic non-small cell lung cancer.
5. Patients with disease previously untreated with systemic therapy must have ≥ 50% PD-L1 staining and patients who have previously received systemic therapy must have ≥ 1% PD-L1 staining on immunohistochemistry
6. Patients must have at least 1-3 lesions suitable for treatment with stereotactic radiotherapy.
7. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumour lesion where feasible. Newly-obtained is defined as a specimen obtained up to 12 weeks prior to randomisation. Patients for whom newly-obtained samples cannot be provided (e.g. inaccessible or patient safety concern) may submit an archived specimen only upon agreement from the study principal investigators.
8. Have a performance status of 0-1 on the ECOG Performance Scale (see Appendix 1).
9. Demonstrate adequate organ function as defined in table 3 below, all screening labs should be performed within 10 days of randomisation.

   Table 3 Adequate Organ Function Laboratory Values

   Absolute neutrophil count (ANC) ≥1.5x109/L Platelets≥100x109L Haemoglobin ≥90 g/L without transfusion or EPO dependency (within 7 days of assessment)

   Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥30 mL/min for patients with creatinine levels > 1.5 X institutional ULN

   Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT)≤ 2.5 X ULN OR ≤ 5 X ULN for patients with liver metastases

   International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants ≤1.5 X ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
10. Life expectancy > 3 months.
11. Be willing and able to comply with all study requirements, including treatment, attending assessments and follow-up.
12. Female patient of childbearing potential should have a negative urine or serum pregnancy within 7 days of randomisation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. Female patients of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (See Section 8.10). Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
14. Male patients should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Has had previous high dose radiotherapy (biological equivalent of >30Gy in 10#) to an area to be treated which includes vertebral bodies (see below).

   Note: Previous high dose radiotherapy is defined as a biological equivalent dose to above that of 30 Gy in 10 fractions using an alpha/beta ratio (50) of 3.

   Where a patient has received radiotherapy to an equivalent or lower dose than defined above, stereotactic radiotherapy of the area may be considered. In doing so, assessment of the volume and total dose received by any overlap region must be made, and documented by generating a cumulative plan incorporating both the previous and current treatment fields. It is the treating radiation oncologist's responsibility to review both the current plan and the cumulative plan inclusive of previous radiotherapy.
2. Has had previous thoracic radiotherapy of > 36Gy within the 6 months prior to randomisation.
3. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with small asymptomatic or previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of enlarging brain metastases, and are not using steroids for intracranial neurological symptoms at least 7 days prior to trial randomisation. This exception does not include leptomeningeal disease which is excluded regardless of clinical stability.
4. Has evidence of Spinal Cord Compression.
5. Has a Spinal Instability Neoplastic Score ≥ 7 unless lesion reviewed by a neurosurgical service and considered stable (see Appendix 2).
6. Requires surgical fixation of bone lesion for stability. All surgical fixation and instrumentation must be completed before randomisation on study.
7. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of randomisation.
8. Has a diagnosis of immunodeficiency.
9. Has a known history of active TB (Bacillus Tuberculosis).
10. Has a hypersensitivity to pembrolizumab or any of its excipients.
11. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to randomisation or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
12. Has diagnosed and/or treated additional malignancy within 5 years prior to randomisation with the exception of: curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, curatively treated early stage cervical cancer, breast cancer or prostate cancer with no evidence of active disease. Other exceptions may be considered following consultation with the principal investigator
13. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
14. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
15. Has had any systemic anti-cancer therapy or radiation therapy within 4 weeks prior to randomisation
16. Has known interstitial lung disease
17. Has an active infection requiring systemic therapy.
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
20. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
21. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
22. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
23. Has received a live vaccine within 30 days of randomisation. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu- Mist®) are live attenuated vaccines, and are not allowed. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: National Cancer Institute CTCAE version 4.03 criteria. — https://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- SABR Plus Pembrolizumab: SABR (18-20Gy) to 1-3 lesions followed 7 (+/-2) days later by pembrolizumab 200mg every 3 weeks for 24 months.
- Pembrolizumab Plus SABR: Pembrolizumab 200mg every 3 weeks for 24 months with SABR (18-20Gy) to 1-3 lesions delivered 7 (+/-2) days after first dose of Pembrolizumab.
Period: Overall Study
Arm/Group | SABR Plus Pembrolizumab | Pembrolizumab Plus SABR
Started | 5 | 8
Completed | 5 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SABR Plus Pembrolizumab | Pembrolizumab Plus SABR | Total
Number analyzed (Participants) | 5 | 8 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (10) | 68 (8) | 66 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 1 | 7 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Measured Using CTCAE Version 4.03
Description: Number of participants with grade 3 treatment related adverse events as determined using CTCAE version 4.03 criteria. Grade 3 treatment-related events are high grade toxicities.
Time Frame: Up to 24 months after commencement of treatment
Measure: Number; unit: participants with G3 TRAEs.
Arm/Group | SABR Plus Pembrolizumab | Pembrolizumab Plus SABR
Number analyzed (Participants) | 5 | 8
participants with G3 TRAEs. | 0 | 1

2. Secondary Outcome: Number of Participants With Overall Response (CR + PR) Assessed Using RECIST 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Assessed up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | SABR Plus Pembrolizumab | Pembrolizumab Plus SABR
Number analyzed (Participants) | 5 | 8
Participants | 4 | 4

3. Secondary Outcome: Number of Participants With Overall Response (irCR + irPR) Assessed Using irRECIST
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (irRECIST) for all lesions and assessed by CT: irComplete Response (CR), Disappearance of all target lesions; irPartial Response (PR), >=30% decrease in TMTB; Overall Response (OR) = irCR + irPR.
Time Frame: Assessed up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | SABR Plus Pembrolizumab | Pembrolizumab Plus SABR
Number analyzed (Participants) | 5 | 8
Participants | 4 | 4

4. Secondary Outcome: Number of Participants With Overall Response (CMR + PMC) Assessed Using PERCIST1.0
Description: Per PERCIST 1.0 Criteria for all lesions and assessed by PET/CT: Complete Metabolic Response (CMR), complete resolution of 18F-FDG uptake; Partial Metabolic Response (PMR), >=30% decrease in target measurable tumour 18F-FDG SUL peak; Overall Response (OR) = CMR + PMR.
Time Frame: Assessed up to 24 months
Population: One patient withdrew consent at cycle 3 from the Pembrolizumab plus SABR Arm, therefore no PET scans were performed and no data available.
Measure: Count of Participants; unit: Participants
Arm/Group | SABR Plus Pembrolizumab | Pembrolizumab Plus SABR
Number analyzed (Participants) | 5 | 7
Participants | 3 | 3

5. Secondary Outcome: Number of Participants With Overall Response (CMRv + PMRv) Assessed Using Peter Mac Metabolic Response Criteria
Description: Per Peter Mac Metabolic Response Criteria In Solid Tumors Criteria (irRECIST) for a lesion and assessed by PET/CT: Complete Metabolic Response (CMRv), FDG activity within tumour site decreased to equal or less than adjacent soft tissue; Partial Metabolic Response (PMRv), any appreciable reduction in intensity of tumour FDG update or in tumour volume; Overall Response (OR) = CMRv + PMRv.
Time Frame: Assessed up to 24 months
Population: One patient withdrew consent at cycle 3 from the Pembrolizumab plus SABR ARM, therefore no PET scans were performed.
Measure: Count of Participants; unit: Participants
Arm/Group | SABR Plus Pembrolizumab | Pembrolizumab Plus SABR
Number analyzed (Participants) | 5 | 7
Participants | 3 | 4

6. Secondary Outcome: Percentage of Participants With Overall Survival
Description: From randomisation until the date of death from any cause assessed up to the date when the last patient has their 24 months assessment
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SABR Plus Pembrolizumab | Pembrolizumab Plus SABR
Number analyzed (Participants) | 5 | 8
percentage of participants | 80 [20 to 97] | 50 [15 to 77]

7. Secondary Outcome: Percentage of Participants With Progression Free Survival (PFS)
Description: From randomisation until the date of first progression or until the date of death from any cause, whichever occurs first, assessed up to the date when the last patient has their 12 months assessment
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SABR Plus Pembrolizumab | Pembrolizumab Plus SABR
Number analyzed (Participants) | 5 | 8
percentage of participants | 60 [13 to 88] | 43 [10 to 73]

ADVERSE EVENTS:
Time Frame: Up to 2 years.
Arm/Group | SABR Plus Pembrolizumab | Pembrolizumab Plus SABR
All-Cause Mortality (participants affected / at risk) | 1/5 | 4/8
Serious Adverse Events (participants affected / at risk) | 2/5 | 3/8
Other Adverse Events (participants affected / at risk) | 0/5 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SABR Plus Pembrolizumab (N=5) | Pembrolizumab Plus SABR (N=8)
Cortical thinning (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (2) | 0
Reaccumulation of pericardial effusion (Cardiac disorders) | 1 (1) | 0
Non ST elevation myocardial infarct (Cardiac disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT03307759/Prot_SAP_000.pdf